CLINICAL TRIAL: NCT06216249
Title: A Phase 2 Randomized Trial in Patients With Metastatic Castration Resistant Prostate Cancer to Determine the Efficacy of a Flexible Dosing Schedule of Lu-PSMA Treatment up to 12 Cycles Including Potential Treatment Holiday Periods in Comparison to the Standard Fixed Dosing Schedule of Six Cycles Every Six Weeks (FLEX-MRT)
Brief Title: Phase 2 Randomized Trial of Flexible Dosing Schedule of 177Lu-PSMA-617 for the Treatment of Metastatic Castration-Resistant Prostate Cancer (FLEX-MRT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-000931; NCI-2023-07172 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-11-30; First posted 2024-01-22 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Prostate Carcinoma; Stage IVB Prostate Cancer American Joint Committee on Cancer (AJCC) v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Pluvicto; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (177Lu-PSMA-617) (Experimental): Patients receive 177Lu-PSMA-617 IV once every 6 weeks on study. Beginning with the third cycle, treatments may be postponed beyond the 6 weeks interval based on defined response criteria ("treatment holiday" period). Treatment repeats every 6 weeks for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients receive 68Ga-PSMA-11 IV and undergo PSMA PET/CT throughout the trial. Patients also undergo SPECT/CT, PET/CT, or CT on the trial.
  Interventions: Procedure: Computed Tomography; Other: Gallium Ga 68 Gozetotide; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Positron Emission Tomography; Procedure: PSMA PET Scan; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography
- Arm II (177Lu-PSMA-617) (Active Comparator): Patients receive 177Lu-PSMA-617 IV once every 6 weeks on study. Treatment repeats every 6 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients receive 68Ga-PSMA-11 IV and undergo PSMA PET/CT throughout the trial. Patients also undergo SPECT/CT, PET/CT, or CT on the trial.
  Interventions: Procedure: Computed Tomography; Other: Gallium Ga 68 Gozetotide; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Positron Emission Tomography; Procedure: PSMA PET Scan; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PSMA PET/CT, SPECT/CT, PET/CT and CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Other: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; AAA 517; AAA-517; AAA517; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Drug: Lutetium Lu 177 Vipivotide Tetraxetan — Given IV
  Other Names: 177Lu-labeled PSMA-617; 177Lu-PSMA-617; AAA 617; AAA-617; AAA617; Lu177-PSMA-617; Lutetium Lu 177-PSMA-617; LUTETIUM LU-177 VIPIVOTIDE TETRAXETAN; Lutetium-177-PSMA-617; Pluvicto
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: PSMA PET Scan — Undergo PSMA PET/CT
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography
Other: Questionnaire Administration — Ancillary studies
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
In advanced metastatic castration resistant prostate cancer (mCRPC) progressing after chemotherapy and androgen receptor (AR)-targeted therapy 177Lu-PSMA-617 is an effective treatment. 177Lu-PSMA-617 RLT is administered with a fixed schedule: 6 treatment cycles, administered every 6 weeks. However, the optimum number of cycles of 177Lu-PSMA in patients who show good response remains unknown. Some patients may benefit from more than 6 cycles of therapy. Additionally, some patients experience a complete or almost complete response before the last cycle. It is unclear whether these patients benefit from the subsequent remaining treatment cycle(s). A treatment holiday period would spare these patients some exposure to the therapy agent and avoid potentially unnecessary toxicity when treatment efficacy is already maximal and additional treatment effect cannot be expected. This randomized phase 2 study compares a group of patients treated with LuPSMA on a flexible and extended dosing schedule including "treatment holiday" periods (investigational arm, up to 12 cycles, as described below) to a control group treated with a fixed dosing schedule of 6 treatments cycles maximum administered every 6 weeks. The flexible dosing schedule in the investigational arm will be based on single photon emission computed tomography (SPECT)/computed tomography (CT) response assessments obtained 24h after injection of LuPSMA therapy cycle. The response assessment during treatment holiday period will be based on positron emission tomography/computed tomography (PET/CT) every 12 weeks. Single-time point SPECT/CT dosimetry protocol at every cycle will be performed and will allow to determine the number of cycles that subjects may receive under the study without exceeding the kidney dose threshold.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess a potential survival benefit (2-year survival rate) of patients treated with Lu 177 vipivotide tetraxetan (177Lu-PSMA-617) therapy on a flexible dosing schedule including up to 12 cycles and potential "treatment holiday" periods in comparison to patients treated with the standard fixed dosing schedule of maximum 6 treatment cycles every 6 weeks.

SECONDARY OBJECTIVES:

I. To determine the safety of the flexible/extended schedule of 177Lu-PSMA-617 therapy.

II. To compare the overall survival (OS) of the flexible/extended schedule of 177Lu-PSMA-617 therapy to the standard-of-care schedule of 177Lu-PSMA-617 therapy.

III. To compare the progression-free survival (PFS) of the flexible/extended schedule of 177Lu-PSMA-617 therapy to the standard-of-care schedule of 177Lu-PSMA-617 therapy.

IV. To compare the disease control rate (DCR) of the flexible/extended schedule of 177Lu-PSMA-617 therapy to the standard-of-care schedule of 177Lu-PSMA-617 therapy.

V. To compare the impact on bone pain level of the flexible/extended schedule of 177Lu-PSMA-617 therapy to the standard-of-care schedule of 177Lu-PSMA-617 therapy.

VI. To compare the impact on health-related quality of life of the flexible/extended schedule of 177Lu-PSMA-617 therapy to the standard-of-care schedule of 177Lu-PSMA-617 therapy.

EXPLORATORY OBJECTIVE:

I. To determine the dosimetry in organs and tumor lesions of the flexible/extended schedule of 177Lu-PSMA-617 therapy.

OUTLINE: Patients are randomized to one of 2 arms.

ARM I: Patients receive 177Lu-PSMA-617 intravenously (IV) once every 6 weeks on study. Treatment repeats every 6 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo post-therapeutic SPECT/CT at every cycle. The flexible dosing schedule in the investigational arm will be based on prostate specific antigen (PSA) and SPECT/CT response assessments obtained 24h after injection of LuPSMA therapy cycle. Based on their response to therapy, patients may be eligible for "treatment holiday" periods. The monitoring during treatment holiday period will be based on PSMA PET/CT every 12 weeks. If disease progresses patients will re-enter the dosing schedule for up to 12 cycles total, every 6 weeks. Patients also receive gallium Ga-68 gozetotide (68Ga-PSMA-11) IV and undergo prostate-specific membrane antigen positron emission tomography/CT (PSMA PET/CT) on the trial.

ARM II: Patients receive 177Lu-PSMA-617 IV once every 6 weeks on study. Treatment repeats every 6 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo post therapeutic SPECT/CT throughout the trial. Patients also receive 68Ga-PSMA-11 IV and undergo PSMA PET/CT on the trial.

Upon completion of study treatment, patients are followed up every 3 months for 24 months from after first cycle of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have prostate cancer proven by histopathology
* Patients must have ≥ 1 metastatic lesion by any imaging (CT, magnetic resonance imaging [MRI], bone scan, PET)
* Patients must have received at least one regimen of chemotherapy for mCRPC
* Patients must have received at least one androgen-receptor signaling inhibitors (ARSI)
* Patients must be eligible by PSMA PET VISION criteria. PSMA PET/CT must be performed within 8 weeks of planned first cycle of 177Lu-PSMA-617
* White blood cell (WBC) ≥ 2,500/ul
* Platelets (PLT) ≥ 100,000/ul
* Hemoglobin (Hb) ≥ 9.0 g/dl
* Absolute neutrophil count (ANC) ≥ 1,500 ul
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patients must be adults ≥ 18 years of age
* Patients must have the ability to understand and sign an approved informed consent form (ICF)
* Patients must have the ability to understand and comply with all protocol requirements

Exclusion Criteria:

* Prior cycle of 177Lu-PSMA-617 therapy
* Less than 6 weeks between last myelosuppressive therapy (including docetaxel, cabazitaxel, strontium-89, samarium-153, rhenium-186, rhenium-188, radium-223, hemi-body irradiation) and first cycle of 177Lu-PSMA-617 therapy
* Glomerular filtration rate (GFR) < 50 ml/min
* Urinary tract obstruction or marked hydronephrosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year survival rate | From the date of the first cycle of Lu 177 vipivotide tetraxetan (177Lu-prostate-specific membrane antigen [PSMA]-617) therapy, up to 2 years
  Will be assessed patients treated with 177Lu-PSMA-617 therapy on a flexible dosing schedule (investigational arm) in comparison to patients treated with the standard fixed dosing schedule of maximum 6 treatments cycles every 6 weeks (control arm). Will be reported using descriptive statistics by means of number and percentage of patients dead 24 months after the first cycle.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 12 cycles and treatment holiday periods, assessed up to 24 months after first cycle of study treatment
  Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE). Descriptive statistics (number and percentage) will be reported separately for adverse events (AE) in total and serious adverse events (SAE) based on CTC. These descriptive statistics will be presented for the whole treatment as well as separate for each cycle. In addition, the relationship of AE to the study drug (related, not related) will be reported. Both results from laboratory test, physical examinations and patients surveys will be included. Distribution of each result will be compared between both groups using appropriate tests (e.g., Mann-Whitney U test).
Overall survival | From the date of the first cycle injection of 177Lu-PSMA-617 until death, assessed up to 24 months after first cycle of study treatment
  Group comparisons performed using appropriate tests including survival analyses (Kaplan-Meier estimator). Descriptive analyses (median, standard deviation) is used.
Progression-free survival (PFS) | The date of the first cycle injection of 177Lu-PSMA-617 to the date of first evidence of progression, or death from any cause, whichever occurs first, assessed up to 24 months after first cycle of study treatment
  Group comparisons performed using appropriate tests including survival analyses (Kaplan-Meier estimator). Descriptive analyses (median, standard deviation) is used. Radiographic progression defined as the date of progression on single photon emission computed tomography (SPECT) by visual increase in tumor volume ≥ 30% compared to baseline ± new sites of disease and/or new sites of prostate-specific membrane antigen (PSMA)-negative disease progression on diagnostic computed to computed tomography (CT) or on PSMA positron emission tomography (PET)/CT. Prostate specific antigen (PSA) progression is the date when a ≥ 25% increase in PSA and an increase of 2 ng/mL or more from the nadir is documented and confirmed by a second consecutive value obtained 3 or more weeks later. Clinical progression defined as marked escalation in cancer related pain, immediate need for initiation of new anticancer treatment, and marked deterioration in Eastern Cooperative Oncology Group (ECOG) performance.
Disease control rate (DCR) | Up to 24 months after first cycle of study treatment
  Will be defined as the proportion of patients achieving radiographic stable disease (SD), partial response (PR) or complete response (CR). CR is defined as absence of PSMA-avid tumor on either imaging modality. On SPECT/CT, PR is defined as a > 30% reduction in visual tumor volume at all sites of involved disease compared to baseline cycle #1, no new sites of PSMA-avid tumor and no new sites of PSMA-negative tumor on diagnostic CT, and SD is defined as no change > 30% in visual tumor volume compared to baseline cycle #1, no new sites of PSMA-avid tumor and no new sites of PSMA-negative tumor on diagnostic CT. Respective response groups on PSMA PET/CT are defined by Response Evaluation Criteria in Prostate-specific membrane antigen PSMA PET/CT criteria. Descriptive analysis will be used to determine the DCR.
DCR by combined radiographic + PSA response | Up to 24 months after first cycle of study treatment
  Will be defined as PSA decline ≥ 50% or radiographic PR/CR as defined above. Descriptive analysis will be used to determine the DCR.
Bone pain level | Up to 24 months after first cycle of study treatment
  Descriptive analysis will be used to evaluate the impact on bone pain level by determining the proportion of patients with pain response defined by improvement from baseline (all patients with ≥ 4/10) of at least 2-point absolute improvement without an overall increase in opiate use.
Performance status | Up to 24 months after first cycle of study treatment
  As measured by Eastern Cooperative Oncology Group (ECOG) performance status scale (minimum 0, maximum 5, with higher scores meaning a worse outcome)
Health related quality of life (pain) | Up to 24 months after first cycle of study treatment
  Will be reported using the Brief Pain Inventory - Short Form patient reported outcome questionnaire (9 questions including scales; minimum 0, maximum 10, with higher scores meaning a worse outcome).
Health related quality of life (major symptoms/toxicities) | Up to 24 months after first cycle of study treatment
  Will be reported using the Functional Assessment of Cancer Therapy - Radionuclide Therapy patient reported outcome questionnaire (15 questions; minimum 0, maximum 5, with higher scores meaning a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States